CLINICAL TRIAL: NCT03978585
Title: Comparison of High Tone Therapy and TENS Therapy in Chemotherapy-induced Polyneuropathy
Brief Title: Comparison of High Tone Therapy and TENS Therapy
Acronym: HIT-CIPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Collaborators: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Robert Sassmann, Principal Inverstigator, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 415-E/2376/7-2018
Record Dates: First submitted 2019-05-27; First posted 2019-06-07 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Nervous System Problem
Keywords: HTEMS; peripheral neuropathy; chemotherapy; TENS therapy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Transcutaneous Electric Nerve Stimulation; Therapeutics

STUDY DESIGN:
Intervention Model Description: The random allocation sequence will be generated using the random number generator available online (www.randomization.com). The unit of randomization will be the individual participant, such that each patient will be randomised to either have use of the HTEMS device (intervention), or TENS device (control intervention). To ensure balance in the sample size across groups, we will perform a stratified block randomisation (ratio 1:1, block size 4). Subjects will be stratified by treatment delivery, taxan and oxaliplatin. To assure concealment of allocation, physicians of the Institute of Physical Medicine and Rehabilitation will report to the Institute of General Practice, Family Medicine and Preventive Medicine as soon as patient recruitment has been completed and then randomisation by computerised sequence generation will be performed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: After baseline data and outcome assessment participants will consecutively be randomly assigned to intervention or control group. Thus, neither patients nor the responsible physician will know about the allocation to the HTEMS or TENS group at the time of recruitment.
  Physicians responsible for the clinical examinations and outcome assessment will be blinded. Due to the technical design of the intervention patients cannot be blinded. The analyst and outcome assessors will be kept blind to patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTEMS Arm (Experimental): High tone therapy (home based) daily for 30 minutes on at least 5 of 7 days per week
  Interventions: Device: high tone external muscle stimulation; Device: transcutaneous electrical nerve stimulation (TENS) therapy
- TENS Arm (Active Comparator): TENS therapy (home based) daily for 30 minutes on at least 5 of 7 days per week
  Interventions: Device: high tone external muscle stimulation; Device: transcutaneous electrical nerve stimulation (TENS) therapy

INTERVENTIONS:
Device: high tone external muscle stimulation — Participants receive self-administered home based high tone therapy for 8 weeks for 30 minutes daily after device instruction
  Other Names: HiTOP 191 therapy device (gbo Medizintechnik, Rimbach, Germany)
Device: transcutaneous electrical nerve stimulation (TENS) therapy — Participants receive self-administered home based TENS therapy for 8 weeks for 30 minutes daily after device instruction
  Other Names: DoloBravo therapy device 10-05 (MTR GmbH, Scheideggweg 7, 12277 Berlin),CE 0123

SUMMARY:
This study evaluates the efficacy of home-based high tone external muscle stimulation (HTEMS) compared to transcutaneous electrical nerve stimulation (TENS) in chemotherapy-induced peripheral neuropathy (CIPN). One half of the participants will receive TENS therapy, the other half will receive High tone external muscle Stimulation. It is expected that HTEMS improves symptoms of CIPN.

DETAILED DESCRIPTION:
One of the most common adverse side effects of chemotherapeutic agents especially in taxanes, platins or vinca alkaloids is chemotherapy-induced peripheral neuropathy (CIPN). Prevalence of CIPN was reported in 30% to 40% of patients treated with neurotoxic chemotherapy and may be transient or permanent. It appears predominantly as sensory neuropathy and affects the peripheral parts of the extremities in a "stocking and glove"-distribution. CIPN often presents with symptoms like paresthesia, pain, numbness or tingling, but motor symptoms can occur as well. Symptoms of CIPN may lead to dose reduction or even early cessation of chemotherapy and therefore may affect overall survival in cancer patients. Currently, no evidence-based treatment (drug or non-drug therapy) is available for CIPN. Several approaches to manage peripheral neuropathy have been proposed, but evidence showing a benefit of these procedures regarding clinically relevant endpoints is scarce. One promising approach to ease CIPN symptoms is the application of electrotherapy. Different types of electrical sensory interventions have been explored in the literature e.g. transcutaneous electrical nerve stimulation (TENS) and high-tone external muscle stimulation (HTEMS).TENS is used in medical settings and in self-administration of patients at home. In TENS only the frequency is modulated. The device sends electrical impulses through conductive rubber electrodes to the skin of the impaired region. The applied frequencies range from 2 to 120 Hertz. The pain region must be in the middle of the two electrodes, which have a maximum distance of 20cm. In contrast to the TENS therapy, the HTEMS operates in-depth directly on the muscle and produces pleasant, but intense and thus effective contractions. Additionally in HTEMS, the amplitude and the frequency are modulated simultaneously. The applied frequencies range continuously from 4096 to 32768 Hertz. Different frequencies activate structures of different size. For this reason, it is important to offer a broad spectrum of frequencies. The electrical stimulation is applied by using conductive rubber electrodes. On the upper limbs as well as on the lower limbs the electrodes are positioned as far as possible proximal and distal. During the treatment the muscle is stimulated to contraction through intervals. One interval consists of three seconds ramp-up time (intensity rises), three seconds holding time (intensity maintains on maximum) and three seconds pause (no stimulation).

The application of HTEMS has been shown to be more effective than TENS in the therapy of diabetic peripheral neuropathy. Furthermore, HTEMS demonstrated improvement in pain, discomfort, sleep disturbance and quality of life in patients with end-stage renal disease due to uremic peripheral neuropathy. So far, little research on HTEMS or TENS in CIPN has been carried out, even if this approach is used in clinical practice. The aim of this study is to evaluate the effect and feasibility of home-based HTEMS in patients with chemotherapy-induced peripheral neuropathy.

This pilot study will be based on a single blinded randomised controlled trial study design with an observation time of eight weeks. Patients with cancer receiving a taxan-or platin-based chemotherapy and symptoms of CIPN will be included. Subjects will be stratified by treatment delivery, taxan and platin. The therapy will start after completed adjuvant chemotherapy after a time period of 4 weeks minimum to exclude patients with spontaneous remission of CIPN and in order to reduce the effect of any known or unknown biases related to the treatment regime. Potential study participants will receive information about the study as soon as symptoms occurred to plan inclusion, randomisation and allocation of appointments. Patients will receive a TENS or HTEMS device after randomisation. Participants who are allocated to the control intervention group will receive TENS therapy. The participant is educated for home-based therapy and the treatment should be used daily for 30 minutes for 8 weeks. Additionally, participants' compliance will be checked by reading out the tool box. Participants are asked to fill out the EORTC CIPN 20 (chemotherapy-induced) and EORTC QLQ-C30 (quality of life) questionnaire at baseline and after 8 weeks. Clinical examination encompassing vibration sensibility, tendon reflexes, temperature sensibility perception of touch and muscel strength will be conducted at the same time points.

The investigators would prefer not to constrain patients to specific daily time points and disturb their individual rhythm. Therefore, the investigators recommend performing the intervention at a regular daily time point adapted to the individual daily routine. The primary endpoint is a change in the EORTC-QLQ-CIPN20 score during the eight weeks of intervention. For our primary endpoint the investigators will use an intention-to-treat analysis according to the CONSORT statement. Furthermore, the investigators will analyse the intensity of intervention (compliance) and the effect on the primary endpoint (for example comparison of infrequently and frequently use of device). A minimum use on 5 of 7days per week is required.

ELIGIBILITY:
* Inclusion criteria:

  * Age 18 years or older
  * Histologically proven cancer
  * ECOG performance score 0-1(Eastern Cooperative Oncology Group)
  * Completed neoadjuvant or adjuvant chemotherapy with taxane or platin
  * Minimum time distance to neurotoxic agent 4 weeks, maximum 24 weeks
  * Clinical diagnosis of CIPN ≥Grade 1 according to CTCAE during or after completion of chemotherapy
  * Ability to complete questionnaires by themselves or with assistance
  * Ability to understand the study regimen, its requirements, risks, and discomforts, and ability and willingness to sign an informed consent form

Exclusion Criteria:

* Ongoing treatment with antitumor treatments with potential neurotoxic side effects (e.g. platins, taxanes, vinca alkaloids, bortezomib or thalidomide)
* Completed chemotherapy with neurotoxic side effects other than taxane or platin
* Pre-existing clinically manifest peripheral neuropathy prior to start of chemotherapy (e.g. caused by radiation or malignant plexopathy, lumbar or cervical radiculopathy, carpal tunnel syndrome, B12 deficiency, AIDS, monoclonal gammopathy, diabetes, heavy metal poisoning amyloidosis, syphilis, hyperthyroidism or hypothyroidism, inherited neuropathy, etc.)
* Peripheral arterial occlusive disease > Grade 1
* Skin conditions such as open sores preventing proper application of the electrodes
* Patients with implantable medical electronic devices (e.g. pace maker, Implantable Cardioverter Defibrillator - ICD, catheter, etc.)
* Patients with myocard damages or cardiac arrhythmia
* Patients with epilepsy
* Patients with febrile illnesses or acute infectious diseases
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of CIPN associated symptoms | 8 weeks
  Improvement of CIPN associated Symptoms will be assessed according to the EORTC CIPN 20 questionnaire.The EORTC QLQ-CIPN 20 contains 20 items assessing sensory (9 items), motor (8 items), and autonomic symptoms (3 items), using a 4-point Likert scale (1 = "not at all," 2 = "a little," 3 = "quite a bit," and 4 = "very much"). All scale scores are linearly converted to a 0-100 scale (0=no sensory impairment, 100=worst sensory impairment)

SECONDARY OUTCOMES:
Assessment of Quality of life | 8 weeks
  The QLQ-C30 Version 3.0 is composed of multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. The functional scales and the symptom scales have four-point scales. These are coded with "Not at all", "A little", "Quite a bit" and "Very much." The global health status includes 2 items and an item range of 6 from "Very bad" to "Excellent". All of the scales and single-item measures range in score from 0 to 100. The principle for scoring is the same in all cases: Estimate the average of the items that contribute to the scale; this is the Raw Score. Use a linear transformation to standardise the Raw Score, so that scores range from 0 to 100. For all scales, the Raw Score is the mean of the component items calculated with a formula included in the manual.
Vibration sensibility | 8 weeks
  Vibration sensibility: is evaluated by the use of a graduated Rydel-Seiffer tuning fork (128Hz) with a scale from 0 to 8. Due to age related neural deconditioning, values ≤4 are considered pathological for patients ≥60 years old, for patients under 60 years old, a score≤5 is regarded as pathological
Tendon reflex | 8 weeks
  Achilles tendon, biceps and patellar tendon reflexes are assessed with a reflex hammer and graded on a 5 point scale of 0 to 4+ with 0 being no response, 1+ being diminished/low normal, 2+ being average/normal, 3+ being brisker than average/possibly indicative of disease, and 4+ being very brisk, hyperactive, with clonus.
Temperature sensibility | 8 weeks
  Is assessed by TipTherm (tip therm Gesellschaft mit beschränkter Haftung, Düsseldorf, Germany). The examiner places the two circular end faces of the instrument alternately and in an irregular sequence on the back of the patient's foot and asks for the sensory impression: cold or less cold? Only correct answers suggest an intact temperature discrimination capability. Incorrect answers or uncertainties are to be understood as temperature sense - disturbance at the investigation site
Perception of touch | 8 weeks
  is evaluated by stroking patients´ upper and lower legs and feet in order to detect reduced or altered sensation due to demyelinisation or axonal degeneration
Assessment of muscle strength | 8 weeks
  Strength of the lower muscles is assessed by asking the patient to perform toe standing/walking and heel standing/walking on both feet (possible, not possible)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Flamm, Prof, Study Director — Paracelsus Medical University
Locations (1):
- Paracelsus Medical University Salzburger Landeskliniken, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briani C, Argyriou AA, Izquierdo C, Velasco R, Campagnolo M, Alberti P, Frigeni B, Cacciavillani M, Bergamo F, Cortinovis D, Cazzaniga M, Bruna J, Cavaletti G, Kalofonos HP. Long-term course of oxaliplatin-induced polyneuropathy: a prospective 2-year follow-up study. J Peripher Nerv Syst. 2014 Dec;19(4):299-306. doi: 10.1111/jns.12097. PMID 25582667
- [Background] Seretny M, Currie GL, Sena ES, Ramnarine S, Grant R, MacLeod MR, Colvin LA, Fallon M. Incidence, prevalence, and predictors of chemotherapy-induced peripheral neuropathy: A systematic review and meta-analysis. Pain. 2014 Dec;155(12):2461-2470. doi: 10.1016/j.pain.2014.09.020. Epub 2014 Sep 23. PMID 25261162
- [Background] Gibson W, Wand BM, Meads C, Catley MJ, O'Connell NE. Transcutaneous electrical nerve stimulation (TENS) for chronic pain - an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2019 Apr 3;4(4):CD011890. doi: 10.1002/14651858.CD011890.pub3. PMID 30941745
- [Background] Humpert PM, Morcos M, Oikonomou D, Schaefer K, Hamann A, Bierhaus A, Schilling T, Nawroth PP. External electric muscle stimulation improves burning sensations and sleeping disturbances in patients with type 2 diabetes and symptomatic neuropathy. Pain Med. 2009 Mar;10(2):413-9. doi: 10.1111/j.1526-4637.2008.00557.x. Epub 2009 Jan 16. PMID 19207234
- [Background] Postma TJ, Aaronson NK, Heimans JJ, Muller MJ, Hildebrand JG, Delattre JY, Hoang-Xuan K, Lanteri-Minet M, Grant R, Huddart R, Moynihan C, Maher J, Lucey R; EORTC Quality of Life Group. The development of an EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy: the QLQ-CIPN20. Eur J Cancer. 2005 May;41(8):1135-9. doi: 10.1016/j.ejca.2005.02.012. Epub 2005 Apr 14. PMID 15911236
- [Derived] Sassmann R, Gampenrieder SP, Rieder F, Johansson T, Rinnerthaler G, Castagnaviz V, Lampl K, Herfert J, Kienberger YT, Flamm M, Schaffler-Schaden D, Greil R. Electrotherapy as treatment for chemotherapy-induced peripheral neuropathy - a randomized controlled trial. Front Neurol. 2024 Dec 24;15:1451456. doi: 10.3389/fneur.2024.1451456. eCollection 2024. PMID 39777312